CLINICAL TRIAL: NCT06105931
Title: Physiologic Markers of Cardiometabolic Risk in People With Type 1 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000036125; 1R01DK134398-01A1 (NIH)
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: type1diabetes; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Young adults with T1D who have a body mass index <25 kg/m2 (Experimental): Young adults with T1D who have a body mass index <25 kg/m2 will have: abdominal MRI, hyperinsulinemic-euglycemic clamp wtih stable isotope tracer, DEXA scan and a High Fat Mixed Meal Tolerance Test.
  Interventions: Biological: Hyperinsulinemic-euglycemic clamp; Other: High Fat Mixed Meal Tolerance Test

INTERVENTIONS:
Biological: Hyperinsulinemic-euglycemic clamp — Hyperinsulinemic-euglycemic clamp will be used to assess insulin resistance. After IVs are placed, participants will be transitioned to intravenous insulin administration for the baseline portion of the study. Stable Isotope Tracer Infusions will assess rates of glucose, lipid metabolism, and beta-hydroxybutyrate turnover during the last 30 minutes of the baseline equilibration period and again during the last 30 minutes of the stepped IV insulin infusion periods.
Other: High Fat Mixed Meal Tolerance Test — After a 12 hour overnight fast, baseline levels of the lipoproteins will be drawn. The YCCI Bionutrition Service kitchen will prepare the standardized high-fat meal. Participants will administer their bolus insulin per their home regimen for the carbohydrates in the high-fat meal, and then they will consume the meal within a 15-minute timeframe.

SUMMARY:
More than 40% of young adults with type 1 diabetes (T1D) also have overweight or obesity. Each of these diagnoses increase the risk of adverse cardiovascular events. Investigators aim to obtain reference data for individuals with T1D who do not have overweight obesity, to understand how close GLP-1 analogue obesity treatment in those with overweight/obesity brings physiologic markers of cardiometabolic risk to those with BMI in the normal range. Specifically, investigators will describe how drivers of gluconeogenesis and lipemia (specifically measured as visceral fat ratio, insulin resistance, and postprandial lipemia,) that contribute to cardiometabolic risk in T1D change over time.

DETAILED DESCRIPTION:
Primary Objective

The primary objectives of this physiologic study are to:

1. examine how visceral adipose tissue (VAT), measured as VAT/Subcutaneous Adipose Tissue + VAT changes over 1 year in young adults with T1D and body mass index <25kg/m2.
2. determine how hepatic insulin resistance changes over 1 year in young adults with T1D and body mass index <25kg/m2.
3. determine how the area under the curve of triglycerides after a high fat mixed meal tolerance test changes over 1 year in young adults with T1D and body mass index <25kg/m2.

Secondary Objective

The secondary objective[s] of this study are to determine change in:

Aim 1: Weight and % body fat from baseline to 1 year. Aim 2: Suppression of endogenous glucose production (a measure of insulin resistance), expressed as the change in endogenous glucose rate of appearance (mg/kg/min) at baseline and during the low dose (hepatic) phase, and relationship to VAT/(VAT+SAT) from baseline to 1 year. Glucose rate of appearance, glycerol rate of appearance, glucose oxidation, and fat oxidation will be assessed in all clamp phases baseline to 1 year.

Aim 3: Postprandial rise in other atherogenic lipoproteins baseline to 1 year. The data obtained from this protocol will serve as reference data for a randomized clinical trial of GLP-1 analogue obesity in young adults with T1D and overweight/obesity.

The focus of this registration is the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 to ≤30 years
* Diagnosed T1D for at least 12 months and with BMI <25 kg/m2.
* HbA1c ≤10%
* Clinical use of continuous glucose monitoring (CGM)
* Any known laboratory safety parameter consistently outside the below extended laboratory ranges in the past year:

  1. Baseline creatinine >1.0mg
  2. Hypertriglyceridemia (>400 mg/dl)
  3. ALT ≥3.5 times the upper normal limit (UNL)

Exclusion Criteria:

* Current use of adjunctive diabetes medication or anti-obesity medication
* Insulin dose <0.5 units/kg/day
* Use of lipid lowering prescription medication other than statins or omega-3 products
* Doesn't meet MRI safety criteria or having claustrophobia
* Known liver disease other than non-alcoholic steatosis or non-alcoholic fatty liver disease
* Known renal impairment
* Pregnancy or lactation, or planning to become pregnant during the study period.
* Anemia or known hematologic condition impacting HbA1c reading, or another medical condition that precludes participation.
* Treatment with another investigational drug within the past 1 month
* Past medical history of or self-reported corn allergy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in VAT/(VAT+SAT) from baseline to 1 year | baseline and 1 year
  Measured as VAT/Subcutaneous Adipose Tissue + VAT changes over 1 year in young adults with T1D and body mass index <25kg/m2.
Change in hepatic insulin resistance from baseline to 1 year | baseline and 1 year
  Hepatic insulin resistance, measured by beta-hydroxybutyrate (surrogate marker of acetyl-CoA, which regulates gluconeogenesis), changes over 1 year in young adults with T1D and body mass index <25kg/m2.
Change in triglycerides from baseline to 1 year | baseline and 1 year
  Change in triglycerides after a high-fat mixed meal tolerance test, expressed as the total Area Under the Curve (AUCTG) over 6 hours from baseline to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Van Name, MD, Principal Investigator — Yale University
Locations (1):
- Yale Pediatric Diabetes Research, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No